CLINICAL TRIAL: NCT05097261
Title: Brain Injury and Ketamine: a Prospective, Randomized Controlled Double Blind Clinical Trial to Study the Effects of Ketamine on Sedative Sparing and Intracranial Pressure in Traumatic Brain Injury Patients.
Brief Title: Ketamine in Acute Brain Injury Patients.
Acronym: BIKe
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Geert Meyfroidt, MD, PhD (Other)
Collaborators: University of Liege (Other); Centre Hospitalier Régional de la Citadelle (Other); AZ Delta (Other); AZ Sint-Jan AV (Other); AZ Turnhout (Other); Imelda Hospital, Bonheiden (Other)
Responsible Party: Sponsor-Investigator, Geert Meyfroidt, MD, PhD, Associate Professor of Medicine, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: S60859; 2017-004698-15 (EudraCT Number)
Record Dates: First submitted 2020-09-08; First posted 2021-10-28 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Racemic ketamine® will be administered by continuous infusion in a prefilled 50 ml syringe at a concentration of 50 mg/ml, undiluted. The ketamine dose is 1 mg/kg/h, to a maximum dose of 120 mg/hour, which corresponds to an infusion rate of 0.02 ml/kg/h to a maximum rate of 2.4 ml/h. Study patients weighing over 120 kg will not exceed the maximum dose of 120mg/kg of ketamine.
  The study medication will be started within 6 hours after randomization. The IMP, ketamine, will be provided directly to each Participating Site by the official supplier of ketamine for Belgium (Pfizer).
  Interventions: Drug: Ketamine
- Placebo (Active Comparator): The placebo (NaCl 0.9%) will be provided in the same type syringes and administered at the same infusion rate as the IMP (0.02 ml/kg/h to a maximum rate of 2.4 ml/h).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Racemic ketamine® will be administered by continuous infusion in a prefilled 50 ml syringe at a concentration of 50 mg/ml, undiluted. The ketamine dose is 1 mg/kg/h, to a maximum dose of 120 mg/hour, which corresponds to an infusion rate of 0.02 ml/kg/h to a maximum rate of 2.4 ml/h.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Placebo — Placebo (NaCl 0.9%) will be provided in the same type syringes and administered at the same infusion rate as the IMP (0.02 ml/kg/h to a maximum rate of 2.4 ml/h).
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Although, in the past years, an increasing use of ketamine in Traumatic Brain injury (TBI) has been reported as an adjunct to other sedatives, there is no evidence from randomized clinical trial to support this practice.

The BIKe (Brain Injury and Ketamine) study is a double-blind placebo controlled randomized multicenter clinical trial to examine the safety and feasibility of using ketamine as an adjunct to a standard sedative strategy in TBI patients.

DETAILED DESCRIPTION:
In this study the effects of ketamine as an adjunct to an standard sedation regime in adult TBI patients will be investigated on the therapy intensity level and intracranial pressure. All patients will receive propofol for sedation to control ICP, to a maximum dose of 4 mg/kg/h. If the ICP is not controlled at the maximum dose of propofol, midazolam will be added, to a maximum dose of 0.3 mg/kg/h, as part of the current standard of care in the Participating Sites. All patients will receive remifentanil, fentanyl or sufentanil infusions for pain relief. The study medication (ketamine or placebo) will be started after randomization.

As part of the current standard of care in the Participating Sites, the decision for decompressive craniectomy and/or barbiturate coma will be taken after multidisciplinary consultation between the treating intensivist and neurosurgeon.

The decision to stop or reduce sedation, lies with the treating physician, based on the level of ICP control, the absence of clinical or radiological signs of deterioration of the neurologic state. In the case of barbiturate coma, the study drug will be discontinued. During and following decompressive craniectomy, the sedative regime (propofol/midazolam/study drug/ opioids) will be continued. In case of suspected or threatening Propofol-Related Infusion syndrome, propofol will be stopped and switched to midazolam. In case of hypertriglyceridemia >200 mg/dL, propofol will be reduced and if necessary, midazolam will be associated to allow control of sedation. During surgical procedures related to the traumatic brain injury or not, the study drug will not be discontinued. The use of open label administration of ketamine is not allowed during the course of the trial, i.e until hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury patients
* Age >= 18 years
* Admitted to the ICU
* Within 72 hours after admission to the initial hospital:

  * ICP monitoring in place (parenchymal probe, ventricular catheter, or both)
  * Requiring sedation

Exclusion Criteria:

* Known pregnancy and/or lactation
* Imminent or actual brain death upon inclusion
* Allergy or intolerance to the study medication
* Pre-existing neurocognitive disorders, pre-existing congenital or non-congenital brain dysfunction.
* Inability to obtain informed consent
* Inclusion in an interventional randomised controlled trial of which the PI indicates that co-inclusion specifically in the BIKe study is prohibited.
* Therapy restriction code upon inclusion.
* Porphyria
* Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in therapeutic intensity of intracranial pressure (ICP) reducing measures, assessed by the TIL score (Therapy Intensity Level) | From date of randomization (and start study drug) until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months.
  The primary efficacy endpoint will be the reduction in daily Therapy Intensity Level (TIL) score, based on the highest score in each item per day until study drug discontinuation (calculated every day on the available data at 7:00 AM). Scales for TIL score range from 0 (minimum) to 38 (maximum). Higher scores are related to worse outcome.

SECONDARY OUTCOMES:
Intracranial pressure (ICP) | From date of randomization until study drug discontinuation or or date of death from any cause, whichever came first, assessed up to 6 months.
  The average of hourly validated intracranial pressure (mmHg) measurements per 24 hours
Duration of sedation | defined as the start of the first infusion of either propofol, midazolam and/or dexmedetomidine to the cessation of the last uninterrupted infusion of either propofol, midazolam, opioids and/or dexmedetomidine, assessed up to 6 months.
  Total duration of the first period of sedative treatments (propofol, midazolam and/or dexmedetomidine)
Propofol | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed at ICU discharge, assessed up to 6 months.
  Total dose of propofol in mg per 24 hours
Mechanical ventilation | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months.
  Total duration of mechanical ventilation, defined as all types of ventilation where positive end expiratory pressure is applied, expressed in cm H2O (5 cm H2O minimum).
Midazolam | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months.
  Total dose of midazolam in mg per 24 hours
ICU length of stay | From ICU admission until ICU discharge (end of stay is defined as application for discharge in the hospital computer system, or death), assessed up to 6 months.
  Length of stay (number of days) in ICU
Hospital length of stay | From admission to hospital until end of stay in hospital (dead or alive), assessed up to 6 months.
  Length of stay in hospital (days)
Richmond Agitation-Sedation scale (RASS) | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months.
  Average daily RASS. Scale ranges from +4 (combative) until -5 (Unarousable).
Delirium | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months.
  Number of delirium-free days, assessed 3 times per day with the Intensive Care Delirium Screening Checklist (ICDSC) or Confusion Assessment Method for the ICU (CAM-ICU delirium scale).
eGOS | 6 months after the onset of TBI
  extended Glasgow Outcome Scale (eGOS)
ICU mortality | From date of randomization until ICU discharge, assessed up to 6 months.
  Mortality during ICU stay
In-hospital mortality | From date of randomization until hospital discharge, assessed up to 6 months.
  Mortality during hospital stay
Barbiturate coma incidence | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months.
  The incidence of barbiturate coma
Barbiturate coma duration | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months.
  The duration of barbiturate coma
Decompressive craniectomy | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months, assessed up to 6 months.
  The incidence of decompressive craniectomy
Propofol Infusion Syndrome (PRIS) | From date of randomization until study drug discontinuation or date of death from any cause, whichever came first, assessed up to 6 months.
  Incidence of PRIS documented and diagnosed by the attending physician and defined as:
  * Cardiac manifestations, not explained by a coronary ischemic event:
    * Acute refractory bradycardia leading to asystole, or
    * ECG: widening of QRS-complex, or Brugada-syndrome-like patterns (particularly Type 1: Coved-type ST-segment elevation >2mm in >1 of V1-V3 followed by a negative T-wave), or ventricular tachy-arrhythmias
  * Combined with one or more of the following:
    * Unexplained metabolic acidosis (base deficit > 10 mmol/L)
    * Rhabdomyolysis (Creatinine kinase at least five times the upper limit of normal)
    * Hyperlipidaemia (triglyceride levels > 150 mg/dl)
    * Enlarged or fatty liver, apparent on CT or echography
  * All occurring in patients receiving propofol for > 24h
  * Diagnosed by the attending physician

CONTACTS AND LOCATIONS:
Overall Officials: Geert Meyfroidt, MD PhD, Principal Investigator — Associate Professor of Medicine
Locations (8):
- Belgium (8):
  - Imelda Bonheiden, Bonheiden
  - AZ Sint-Jan, Bruges
  - Jessa Ziekenhuis, Hasselt
  - UZLeuven, Leuven
  - CHR de la Citadelle Liège, Liège
  - CHU de Liège, Liège
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Sloovere V, Mebis L, Wouters P, Guiza F, Boonen E, Bourgeois M, Dubois J, Ledoux D, Lormans P, Marechal H, Van der Hauwaert E, Depreitere B, Meyfroidt G. Brain Injury and Ketamine study (BIKe): a prospective, randomized controlled double blind clinical trial to study the effects of ketamine on therapy intensity level and intracranial pressure in severe traumatic brain injury patients. Trials. 2025 May 28;26(1):177. doi: 10.1186/s13063-025-08835-5. PMID 40437634